CLINICAL TRIAL: NCT04459845
Title: Early Intervention For Families Experiencing Homelessness: A Randomized Trial Comparing Two Parenting Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Lotus House (Unknown)
Responsible Party: Principal Investigator, Paulo A. Graziano, PhD, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-17-0265-CR02
Record Dates: First submitted 2020-06-18; First posted 2020-07-07 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Behavior Problem; Parenting
Keywords: early intervention; parenting; homelessness; parent child interaction therapy; child parent psychotherapy; behavior problems; trauma symptoms
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor are masked to the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Child Interaction Therapy (Active Comparator): Parents and children will receive 12 weekly sessions of PCIT.
  Interventions: Behavioral: Parent Child Interaction Therapy
- Child Parent Psychotherapy (Active Comparator): Parents and children will receive 12 weekly sessions of CPP
  Interventions: Behavioral: Child Parent Psychotherapy

INTERVENTIONS:
Behavioral: Parent Child Interaction Therapy — Parent-child Interaction therapy (PCIT; Eyberg and Robinson, 1982) s a manualized evidence-based behavioral parent training program that integrates social learning and attachment theories. Parents proceed through two distinct phases: Child-Directed Interaction (CDI) resembles traditional play therapy, and Parent-Directed Interaction (PDI) resembles clinical behavior therapy. During all sessions, the therapist coaches each parent in vivo in their use of the CDI and PDI skills with their child.
  Arms: Parent Child Interaction Therapy
Behavioral: Child Parent Psychotherapy — Child-parent psychotherapy (CPP; Lieberman et al., 2005) is a relationship-based treatment that integrates attachment, cognitive-behavioral, social-learning, and psychodynamic theories. CPP focuses on the child-parent relationship as a way to improve the child's adaptive functioning. Various treatment strategies are employed including a focus on safety, affect regulation, the joint construction of a trauma narrative, and engagement in developmentally appropriate activities.
  Arms: Child Parent Psychotherapy

SUMMARY:
This study aims to compare the efficacy in delivering two evidence-based parenting programs to families and young children experiencing homelessness. Outcomes evaluated include feasibility, treatment completion, treatment satisfaction of delivery of interventions as well as child outcomes (e.g., behavior problems, trauma symptoms) and parenting outcomes (parenting stress and parenting skills).

DETAILED DESCRIPTION:
The number of homeless families in the U.S. has increased since the 1980s to over half a million as of 2018. Most troubling, in 2013 (the most recent year for which census data is available) one in every 30 children in the U.S., or 2.5 million, experienced homelessness. In addition to having disproportionally higher rates of unmet health needs (e.g., acute health problems, trauma-related injuries), children experiencing homelessness have staggering mental health needs such that 78% suffer from at least one mental health issue (e.g., depression, behavior problems) along with academic/developmental delays. Given that over half of all homeless children in the US are under the age of 6, it is particularly important to investigate the effectiveness of evidence-based parenting programs within a homeless population. This study aims to compare the efficacy in delivering two evidence-based parenting programs to families and young children experiencing homelessness.

ELIGIBILITY:
Inclusion Criteria:

* Any child between the ages of 2 and 5 and his/her mother who is currently homeless and living in the Lotus House shelter.

Exclusion Criteria:

* Family is already involved in a parenting program or does not speak English or Spanish.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory (ECBI) | 16 weeks after start of intervention
  Change in overall externalizing behavior problems
Child and Adolescent Trauma Screener (CATS) | 16 weeks after start of intervention
  Change in overall PTSD symptom severity
Parenting Stress Index Short Form 4th edition (PSI-SF) | 16 weeks after start of intervention
  Change in overall level of parenting stress
The Dyadic Parent-Child Interaction Coding System | 16 weeks after start of intervention
  Change in positive and negative parenting skills observed during 5 minute child led play session

SECONDARY OUTCOMES:
Therapy Attitude Inventory | 16 weeks after start of intervention
  Mothers' satisfaction with treatment
Treatment Attendance | 16 weeks after start of intervention
  Percentage of families who completed the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Graziano, Ph.D, Principal Investigator — Florida International University
Locations (1):
- Lotus House, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified summary data from the study will be shared with other researchers upon request and after completion of study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of study and for 3 years.

REFERENCES:
- [Derived] Graziano PA, Spiegel JA, Hayes T, Arcia E; Sundari Foundation. Early intervention for families experiencing homelessness: A pilot randomized trial comparing two parenting programs. J Consult Clin Psychol. 2023 Apr;91(4):192-207. doi: 10.1037/ccp0000810. PMID 37166851